CLINICAL TRIAL: NCT02431390
Title: Effect of RAPAELⓇ Smart Glove Digital Treatment System on Upper Limb Functional Recovery and Brain Plasticity in Stroke Patients
Brief Title: Upper Limb Biofeedback Rehabilitation System (RAPAELⓇ Smart Glove Digital Treatment System) Training for Stroke Recovery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pusan National University (Other)
Collaborators: Samsung Medical Center (Other); Sungkyunkwan University (Other); NEOFECT Rehabilitation Solutions (Other)
Responsible Party: Principal Investigator, Yong-il Shin, Associate Professor, Pusan National University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PNUYH-03-2015-002
Record Dates: First submitted 2015-04-12; First posted 2015-05-01 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Stroke; Cerebral Vascular Accident
Keywords: RAPAELⓇ Smart Glove digital treatment system; Rehabilitation; Stroke; Upper limbs
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RAPAELⓇ Smart Glove group (Experimental): The experimental group includes 40 stroke patients. The group will receive the conventional occupational therapy(30min per session, 5 times per week, during 4 weeks of hand dexterity training) and RAPAELⓇ Smart Glove digital treatment system training. RAPAELⓇ Smart Glove digital treatment training will consist of games and play to facilitate the function of upper limbs and brain plasticity. RAPAELⓇ Smart Glove group will be provided the 20 training session. (30min per session, 5 times per week, during 4 weeks)
  Interventions: Device: RAPAELⓇ Smart Glove digital treatment system
- Additional occupation therapy group (Active Comparator): The active comparator group includes 40 stroke patients.The occupational therapy group will receive the conventional occupational therapy(30min per session, 5 times per week, during 4 weeks of hand dexterity training) sessions twice. Additional conventional occupational therapy sessions are comprised of the training for upper limb and cognition. The additional occupational therapy group will be provided the 20 additional session (30min per session, 5 times per week, during 4 weeks)
  Interventions: Behavioral: Additional occupational therapy

INTERVENTIONS:
Device: RAPAELⓇ Smart Glove digital treatment system — The RAPAELⓇ Smart Glove digital treatment system is constituted for stroke rehabilitation. For use, stroke patients wear the gloves and play the games or puzzle for rehabilitation of upper limbs. The system provides biofeedback to user.
  Arms: RAPAELⓇ Smart Glove group
Behavioral: Additional occupational therapy — 30 minutes of additional conventional occupational therapy session composed of hand dexteriy training
  Arms: Additional occupation therapy group

SUMMARY:
This study is to investigate whether the RAPAELⓇ Smart Glove digital treatment system improves the upper extremity function of stroke patients compared to other clinical treatment by measuring serial behavioral and neuroimaging assessments and to find out therapeutic effect or adverse effect and patient's feed back responses

DETAILED DESCRIPTION:
80 stroke patients(subacute=40, chronic=40) were recruited and randomized to receive either occupation therapy(OT) with or without RAPAELⓇ Smart Glove digital therapy. Groups were divided as follow: Group 1 (5times/4wks, total 20 sessions) Conventional occupation therapy + additional occupation therapy(30min). Group 2 (5times/4wks, total 20 sessions) Conventional occupation therapy + RAPAELⓇ Smart Glove digital treatment(30min).

After the baseline assessment, patients are divided into two groups by drawing for simple random sampling. Total four times of behavioral and neuroimaging assessments were evaluated at baseline, immediately and 2 weeks after each 10 sessions and at 4 weeks after the final session. Assessment tools are as follow:

1. Primary outcome.

   -Fugl-Meyer assessment,
2. Motor and sensory function. MMT&ROM, Motricity index(MI),Action Research Arm test(ARAT), Box&block test, Box&Block test, 9-hole pegboard test, Jebsen-Taylor hand function test, Modified Ashworth scale(MAS), Grip strength test, Grasp/pinch power, Visual analogue scale(VAS), Sensory test(two point discrimination, monofilament)
3. Activity of daily living. Korean version of Modified Barthel index (K-MBI)
4. Cognition function test. Korean-mini mental state examination (K-MMSE)
5. Depressive mood. Korean-Geriatric Depression Scale (K-GDS)
6. Quality of life. Short form-8(SF-8)
7. Neuroimaging tools. Motor evoked potentials (MEP), Functional Magnetic Resonance Imaging (fMRI), Functional near-infrared spectroscopy (fNIRS).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who hemiplegic due to stroke
* Subjects who have more than 22 points of Fugl-Meyer Assessment score in upper extremity
* 40 subjects who have diagnosed as stroke before 3weeks to 3 months(subacute)
* 40 subjects who have diagnosed as stroke more than 6 months ago(chronic)

Exclusion Criteria:

* Subjects who have spasticity and upper extremity dysfunction at unaffected side
* Subjects who have bilateral or multiple brain lesion
* Subjects who have non-controllable medial or surgical disease
* Subjects who is less than 20 years old
* Subjects who have pre-existing and active major neurological or psychiatric disease
* Subjects who have less than 10 degrees of active wrist range of motion
* Subjects who can not complete outcome measurement task
* Subjects who have limitation of communication due to aphasia
* Subjects who have less than 17 points of K-MMSE
* Subjects who is pregnant
* Subjects who have pain or other muscle wasting disease which may interrupt upper extremity exercise

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Change in upper extremity function (FMA) | 2 weeks
  Fugl-Meyer Assessment(FMA) of upper extremity

SECONDARY OUTCOMES:
Change in brain plasticity (fMRI) | baseline and 4 weeks and 8 weeks
  fMRI
Change in brain plasticity (fNIRS) | baseline and 4 weeks and 8 weeks
  Functional near-infrared spectroscopy(fNIRS)
Change in upper extremity function (MEP) | baseline and 4 weeks and 8 weeks
  Measured by Motor evoked potential(MEP)
Change in upper extremity function(MMT&ROM) | baseline and 2,4,8 weeks
  Measured by manual muscle test(MMT) & range of motion(ROM)
Change in activities of daily livings (MI) | baseline and 2,4,8 weeks
  Motricity index(MI)
Change in upper extremity function (ARAT) | baseline and 2,4,8 weeks
  Action Research Arm test(ARAT)
Change in upper extremity function (Box&Block test) | baseline and 2,4,8 weeks
  Box&Block test
Change in upper extremity function (9-hole pegboard test) | baseline and 2,4,8 weeks
  9-hole pegboard test
Change in upper extremity function (Jebson-Taylor Hand Function Test) | baseline and 2,4,8 weeks
  Jebson-Taylor Hand Function Test
Change in upper extremity function (Modified Ashworth scale) | baseline and 2,4,8 weeks
  Modified Ashworth scale
Change in upper extremity function (Grip strength test) | baseline and 2,4,8 weeks
  Grip strength test
Change in upper extremity function (Grasp/Pinch power) | baseline and 2,4,8 weeks
  Grasp/Pinch power
Change in upper extremity sensory function (VAS) | from baseline to 2 weeks after each 10 session and 4 weeks after final the session
  Visual Analogue Scale(VAS)
Change in upper extremity sensory function (Two point discrimination and Monofilament) | baseline and 2,4,8 weeks
  Two point discrimination and Monofilament
Change in activities of daily livings (K-MBI) | baseline and 2,4,8 weeks
  Korean version of Modified Barthel index(K-MBI)
Change in cognition function (K-MMSE) | baseline and 2,4,8 weeks
  Korean-mini mental state examination(K-MMSE)
Change in depressive mood (K-GDS) | baseline and 2,4,8 weeks
  Korean-Geriatric Depression Scale(K-GDS)
Change in quality of life (SF-8) | baseline and 2,4,8 weeks
  Short form-8(SF-8)
Change in upper extremity function (FMA) | baseline and 2,4,8 weeks
  Fugl-Meyer Assessment(FMA) of upper extremity

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Il Shin, Ph.D., Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, South Korea